CLINICAL TRIAL: NCT00577707
Title: A Phase II Study of Erlotinib and Chemotherapy for Patients With Stage IB-IIIA NSCLC With EGFR Mutations (ECON)
Brief Title: Erlotinib and Chemotherapy for Patients With Stage IB-IIIA NSCLC With EGFR Mutations (ECON)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-103; NCT00602238 (obsolete NCT alias)
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: Lung Cancer; Erlotinib; clinical stage IB-IIIA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Pemetrexed; Cisplatin

ARMS (1):
- Patients With Stage IB-IIIA NSCLC With EGFR Mutations (Experimental): This is a open label, single center, phase II trial for patients with clinical stage IB-IIIA NSCLC (T1-3N0-2M0) who have resectable tumors that harbor EGFR activating mutations. Patients will receive erlotinib x 3 weeks prior to initiation of concurrent erlotinib and chemotherapy.
  Interventions: Drug: erlotinib; Drug: Pemetrexed; Drug: Cisplatin; Procedure: Resection

INTERVENTIONS:
Drug: erlotinib — One tablet daily of erlotinib pills (150 mg daily) for the first 21 days. After surgery, you will be asked to take adjuvant erlotinib 150 mg po daily x 2 years.
Drug: Pemetrexed — pemetrexed 500 mg/m^2 every 3 weeks for 4 cycles treatment) on the first day of each cycle of treatment.
Drug: Cisplatin — cisplatin 75 mg/m^2 every 3 weeks for 4 cycles treatment) on the first day of each cycle of treatment.
Procedure: Resection

SUMMARY:
The purpose of this study is to try to improve the odds that your cancer may be cured. Pemetrexed and cisplatin are traditional chemotherapy drugs that have been shown to help some patients with non-small cell lung cancer. Many different types of cancer cells, including your type of lung cancer, have a protein on their surface called the epidermal growth factor receptor (EGFR). Stimulation of these receptors can result in growth of cancer cells and progression of cancer. In addition, your cancer has an EGFR mutation (a specific abnormality in the genetic code for EGFR). Erlotinib (TarcevaTM) is a newer drug which has shown benefit for patients with lung cancers that contain an EGFR mutation. Erlotinib works by blocking this receptor and depriving the cancer cells of this message to grow and multiply. In this research study, we plan to combine erlotinib with traditional chemotherapy drugs to see if the combination works better than chemotherapy alone.

The main purpose of this research is to find out the good and bad effects that the combination of these 3 drugs (pemetrexed, cisplatin and erlotinib) has when given to patients with early stage non-small cell lung cancer before surgery. A secondary purpose is to find out the good and bad effects that occur when erlotinib is given to patients after surgery for 2 years.

DETAILED DESCRIPTION:
Chemotherapy and surgery in combination represents the standard of care for patients with resectable stage IB-IIIA NSCLC. However, the 5-year survival continues to be disappointing despite this standard of care. This study incorporates targeted therapy with an epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI) as part of a multimodality strategy for stage IB-IIIA resectable NSCLC tumors with a known EGFR activating mutation. The rationale for including only patients with EGFR mutations is based on recent data that reported that patients with advanced NSCLC whose tumor harbor EGFR activating mutations had an objective response rate of 71% with gefitinib compared with a 1% objective response rate in patients with EGFR wild-type tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of NSCLC
* Patients must have previously untreated stage IB-IIIA NSCLC (T1-3N0-2M0)
* Patients must have lung cancer with a documented EGFR activating mutation (exon 19 deletion, L858R, L861Q)
* Patients must be candidates for resection with curative intent
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded on CT)
* Age greater or equal to 18 years
* Karnofsky performance status greater or equal to 70%
* Normal marrow function: leukocytes greater than or equal to 3,000/μl, absolute neutrophil count greater than or equal to 1,500/μl, platelets greater than or equal to 100,000/μl, hemoglobin greater than or equal to 9 gm/dl
* Adequate renal function, with creatinine less than or equal to 1.3 mg/dl or calculated creatinine clearance greater to or equal to 60ml/min by Cockroft and Gault equation using parameters of age, weight (kg), and baseline serum creatinine (mg/dl)
* Adequate hepatic function: Total bilirubin within normal limits, AST < 1.5 X UNL, alkaline phosphatase < 1.5 X UNL
* Women of childbearing age must have a negative urine or blood pregnancy test
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter
* Patients must have ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior chemotherapy or radiation therapy, with the exception of chemotherapy for nononcologic conditions (ie, methotrexate for the treatment of rheumatoid arthritis)
* Prior treatment with gefitinib, erlotinib, or other drugs that target EGFR
* Patients must not be receiving any other investigational agents
* Any evidence of interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded)
* Patients who report a hearing deficit at baseline, even if it does not require a hearing aid or intervention, or interfere with activities of daily life (CTCAE grade 2 or higher)
* Peripheral neuropathy > grade 1
* Known HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with the study drugs.
* Other serious illness or medical condition including unstable cardiac disease requiring treatment, history of significant neurologic or psychiatric disorders (including psychotic disorders, dementia, or seizures), or active uncontrolled infection
* Women who are pregnant or breast-feeding
* Psychiatric illness or social situation that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Stage IB-IIIA NSCLC With EGFR Mutations: Phase II Study of Erlotinib and Chemotherapy for Patients with Stage IB-IIIA NSCLC with EGFR Mutations
Period: Overall Study
Arm/Group | Patients With Stage IB-IIIA NSCLC With EGFR Mutations
Started | 9
Completed | 6
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Stage IB-IIIA NSCLC With EGFR Mutations
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathologic Complete Response Rate
Description: Complete Response (CR): Disappearance of all clinical evidence of tumor. Partial Response (PR): A 50% or greater decrease in the sum of the products of measured lesions. No simultaneous increase in the size of any lesion or the appearance of new lesions may occur. Non-measurable lesions must remain stable or regress for this category. Minor Response (MR): A > 25% and < 50% decrease in the sum of the products of measured lesions. No simultaneous increase in the size of any lesion or the appearance of new lesions may occur. Non-measurable lesions must remain stable or regress for this category. Stable Disease (SD): A less than 25% decrease. This includes a decrease of less than 25% in the sum of the products of the measured lesions, and any increase of less than 25% in the sum of the products of the measured lesions. There may be no appearance of new disease sites for this category. Progressive Disease (PD): A ≥25% increase in one or more lesions, or appearance of new lesions.
Time Frame: Patients will undergo a CT scan of chest every 3 months for year 1 and every 4 months for year 2. In years 3 and 4, a chest CT or chest x-ray every 6 months.
Measure: Number; unit: participants
Arm/Group | Patients With Stage IB-IIIA NSCLC With EGFR Mutations
Number analyzed (Participants) | 6
participants
  Minor Response (MR) | 1
  Partial Response (PR) | 1
  Stable Disease (SD) | 2
  Progressive Disease (POD) | 2

2. Secondary Outcome: Number of Participants With Response After 21 Days of Single Agent Erlotinib for Stage IB-IIIA NSCLC With a Known EGFR Mutation
Time Frame: calculate the response rate after 21 days of single agent erlotinib
Population: Data was not collected because of lack of accrual.
Arm/Group | Patients With Stage IB-IIIA NSCLC With EGFR Mutations
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With a Response Rate, 3-year Overall Survival and Median Survival of Patients With a Known EGFR Mutation Receiving Neoadjuvant Chemotherapy and Erlotinib (and Adjuvant Erlotinib).
Time Frame: 3 years
Population: Data was not collected because of lack of accrual.
Arm/Group | Patients With Stage IB-IIIA NSCLC With EGFR Mutations
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Patients With Stage IB-IIIA NSCLC With EGFR Mutations
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Stage IB-IIIA NSCLC With EGFR Mutations (N=6)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Stage IB-IIIA NSCLC With EGFR Mutations (N=6)
ALT, SGPT (Blood and lymphatic system disorders) | 1 (1)
AST, SGOT (Blood and lymphatic system disorders) | 1 (1)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Creatinine (Blood and lymphatic system disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (5)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Clin exam)- Oral cavity (General disorders) | 2 (2)
Nausea (General disorders) | 1 (2)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Sweating (diaphoresis) (General disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Analysis was not done on the secondary outcomes because of lack of accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes